CLINICAL TRIAL: NCT00716248
Title: The Bucillamine Study of Holding Remission After Infliximab Dose-off in Patients With Rheumatoid Arthritis Receiving Methotrexate
Brief Title: Bucillamine Study of Holding Remission After Infliximab Dose-off
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saitama Medical University (Other)
Collaborators: Keio University (Other)
Responsible Party: Hideto Kameda, Department of Internal Medicine, School of Medicine, Keio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMC-94
Record Dates: First submitted 2008-07-08; First posted 2008-07-16 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2009-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — bucillamine; Methotrexate

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bucillamine; Drug: methotrexate
- 2 (Active Comparator)
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: bucillamine — bucillamine 100 mg, twice a day
  Arms: 1
Drug: methotrexate — methotrexate 6 mg or more per week

SUMMARY:
Patients with rheumatoid arthritis who have been well controlled with methotrexate plus infliximab may remain in remission or low disease activity without infliximab. And the chance of sustained remission increase by the addition of another DMARD, bucillamine, at the time of discontinuing infliximab. The BuSHIDO trial is the prospective, randomized, controlled study comparing MTX monotherapy and MTX plus bucillamine combination therapy as to the rate of disease flare after discontinuing infliximab.

ELIGIBILITY:
Inclusion Criteria:

* RA according to American College of Radiology (ACR) classification criteria
* Age of 20 or greater
* DAS28-ESR < 3.2 or DAS28-CRP < 2.6 for more than 6 months

Exclusion Criteria:

* Previously teated with bucillamine
* Pregnancy or lactation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The rate of disease flare | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology/Clinical Immunology, Saitama Medical Center, Saitama Medical University, Kawagoe, Saitama, Japan